CLINICAL TRIAL: NCT05878509
Title: Reliability and Validity of the Tampa Scale for Kinesiophobia in Patients With Traumatic Hand-forearm Injuries
Brief Title: Reliability and Validity of the Tampa Scale for Kinesiophobia
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, UMUT ERASLAN, Assistant Professor, Pamukkale University
Other Study IDs: 60116787-020/81396
Record Dates: First submitted 2023-05-08; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Hand Injuries; Forearm Injuries; Trauma
Keywords: hand injuries; forearm injuries; kinesiophobia; psychometrics
MeSH Terms: conditions — Hand Injuries; Forearm Injuries; Wounds and Injuries; Kinesiophobia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with traumatic hand-forearm injuries: The patients between the ages of 18-65 who were referred to the hand rehabilitation unit due to traumatic hand and forearm injuries, those who did not have any neurological, orthopedic, rheumatological disease or surgery history in the relevant extremity and those who did not have communication problems were eligible to participate in the study.
  Interventions: Other: conducting questionnaires; Other: assesment of the severity and pain

INTERVENTIONS:
Other: conducting questionnaires — The patients were administered TSK, Pain Catastrophizing Scale (PCS), Beck Anxiety Inventory (BAI) by face to face interview technique.
Other: assesment of the severity and pain — The Modified Hand Injury Scoring System (MHISS) to determine the severity of the injury, and Visual Analog Scale (VAS) to evaluate perceived pain levels were used.

SUMMARY:
The aim of this study was to investigate the validity and reliability of the Tampa Scale for Kinesiophobia (TSK) in patients with traumatic hand and forearm injuries.

A total of 170 patients with traumatic hand-forearm injuries with a mean age of 37.57±11.85 (18-63) years were included in the study. TSK, Pain Catastrophizing Scale (PCS) and Beck Anxiety Inventory (BAI) were applied to the patients in the first session. Tampa Scale for Kinesiophobia was re-administered 15 days after the first session. Test-retest reliability, internal consistency, and construct validity of the TSK were evaluated. In addition, exploratory factor analysis was applied.

ELIGIBILITY:
Inclusion Criteria:

* patients who had traumatic hand and forearm injuries
* being 18-65 years old

Exclusion Criteria:

* patients who have neurological, orthopedic, rheumatological disease or surgery history in the relevant extremity
* patients who have communication problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients between the ages of 18-65 who were referred to the hand rehabilitation unit due to traumatic hand and forearm injuries, those who did not have any neurological, orthopedic, rheumatological disease or surgery history in the relevant extremity and those who did not have communication problems were eligible to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Tampa Scale for Kinesiophobia (change) | The evaluation were completed in the first session when the patient applied to the hand rehabilitation unit, and it was also repeated 15 days after the first session. The exact time is post-operative/post-injury 2nd week and 4th week. Change
  TSK was developed in 1991 (Miller, Kori, & Todd, 1991), but was not published until 1995 (Liu et al., 2021). It is a 17-item scale and is scored with a 4-point Likert scale (1= Strongly disagree, 4= Strongly agree). A total score ranging from 17 to 68 was obtained after reversing items 4, 8, 12 and 16. The higher the score, the higher the kinesiophobia degree. The Turkish version of the questionnaire has been developed (Yilmaz, Yakut, Uygur, & Uluğ, 2011). The cut-off score of the TSK has been reported as 37 (Wertli, Rasmussen-Barr, Weiser, Bachmann, & Brunner, 2014).
Pain Catastrophizing Scale | The evaluation were completed in the first session for once when the patient applied to the hand rehabilitation unit. The exact time is post-operative/post-injury 2nd week.
  PCS is a scale developed to determine the catastrophic thoughts or feelings about pain experience and ineffective coping skills (Sullivan, Bishop, & Pivik, 1995). It consists of 13 items and three sub-factors: helplessness, magnification and rumination. A Likert-type scale scored between 0-4 is used to obtain a total score ranging from 0 to 52. High score indicates that patients' catastrophizing levels are also high. The Turkish validity-reliability study of the questionnaire was conducted (Ugurlu, Karakas Ugurlu, Erten, & Caykoylu, 2017).
Beck Anxiety Inventory | The evaluation were completed in the first session for once when the patient applied to the hand rehabilitation unit. The exact time is post-operative/post-injury 2nd week.
  BAI is a self-report scale developed by Beck et al. and used to determine the frequency of anxiety symptoms (Beck, Epstein, Brown, & Steer, 1988). It is a Likert-type scale consisting of 21 items each scored between 0 and 3. Turkish validity and reliability were performed by Ulusoy et al (Ulusoy, Sahin, & Erkmen, 1998).

SECONDARY OUTCOMES:
Modified Hand Injury Scoring System | The evaluation were completed in the first session for once when the patient applied to the hand rehabilitation unit.The exact time is post-operative/post-injury 2nd week.
  MHISS is a scoring system developed to determine injury severity in hand and forearm injuries in 4 components: integument (skin and nail), skeletal (bone and ligament), motor (tendon) and neurovascular (nerve and vascular). Each component includes absolute scores and weighted scores considering the functional importance of the affected ray. If there are additional factors such as wound contamination, a compound fracture, crush, or avulsion, the total score for each component is doubled. All anatomical structures missing due to amputation are scored as damaged. The total MHISS is obtained by summing up the scores of all components and divided into four categories as minor (<20), moderate (21-50), severe (51-100) and major (> 101) injuries (Urso-Baiarda et al., 2008).
Visual Analogue Scale | The evaluation were completed in the first session for once when the patient applied to the hand rehabilitation unit.The exact time is post-operative/post-injury 2nd week.
  The pain severity of the patients was evaluated using the Visual Analogue Scale (VAS). "0" indicates no pain, and "10" indicates the most severe pain perceived. Perceived pain levels were questioned during sleeping, resting and activity.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Kitiş, Professor, Study Chair — Pamukkale University Faculty of Physiotherapy and Rehabilitation
Locations (1):
- Pamukkale University, Denizli, Kınıklı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data is available to other researchers upon request.

REFERENCES:
- [Background] Miller RP, Kori SH, Todd DD. The Tampa Scale: a Measure of Kinisophobia. The Clinical Journal of Pain.1991;7(1).
- [Background] LUNDBERG MKE, STYF Jorma, CARLSSON SG. A psychometric evaluation of the Tampa Scale for Kinesiophobia-from a physiotherapeutic perspective. Physiotherapy theory and practice. 2004; 20(2): 121-133.